CLINICAL TRIAL: NCT02532036
Title: A Phase I Trial to Compare the Safety and Immunogenicity of Candidate TB Vaccine MVA85A Administered by the Aerosol Inhaled Route and the Intramuscular Route in Healthy Adult Volunteers Who Are Latently Infected With Mycobacterium Tuberculosis
Brief Title: MVA85A Aerosol vs Intramuscular Vaccination in Adults With Latent Mycobacterium Tuberculosis (M. tb) Infection
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: University of Oxford (Other)
Collaborators: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: TB040
Record Dates: First submitted 2015-08-18; First posted 2015-08-25 (Estimated); Results first posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2018-11

CONDITIONS: Tuberculosis
Keywords: MVA85A; Tuberculosis; Vaccine; Aerosol
MeSH Terms: conditions — Tuberculosis | interventions — MVA 85A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Starter Group (Experimental): Receive 1x10^7 pfu aerosol inhaled MVA85A at day 0.
  Interventions: Biological: Aerosol inhaled MVA85A
- Group A (Experimental): Receive 5x10^7 pfu aerosol inhaled MVA85A, and intramuscular saline placebo both at day 0.
  Interventions: Biological: Aerosol inhaled MVA85A; Biological: Intramuscular Saline placebo
- Group B (Experimental): Receive 5x10^7 pfu intramuscular MVA85A, and aerosol inhaled saline placebo both at day 0.
  Interventions: Biological: Intramuscular MVA85A; Biological: Aerosol inhaled Saline placebo

INTERVENTIONS:
Biological: Aerosol inhaled MVA85A
  Other Names: MVA85A
  Arms: Group A; Starter Group
Biological: Intramuscular MVA85A
  Other Names: MVA85A
  Arms: Group B
Biological: Intramuscular Saline placebo
  Other Names: Saline
  Arms: Group A
Biological: Aerosol inhaled Saline placebo
  Other Names: Saline
  Arms: Group B

SUMMARY:
TB040 is a clinical trial to investigate and compare the effects of a candidate Tuberculosis (TB) vaccine, MVA85A, administered by the aerosol inhaled route and the intramuscular route in healthy adult volunteers who are latently infected with Mycobacterium tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

Volunteers must meet all of the following criteria to enter the trial:

* Healthy adult aged 18-55 years
* Resident in or near Oxford, Birmingham or London for the duration of the trial period
* Screening IGRA positive
* Ineligible for chemoprophylaxis for latent M.tb infection, declined prophylaxis or considered low risk due to distant contact history
* Chest Computed Tomography (CT) normal; or abnormal with features consistent with primary M.tb infection but no features suggestive of active disease
* No relevant findings in medical history or on physical examination
* Allow the Investigators to discuss the individual's medical history with their General Practitioner
* Use effective contraception for the duration of the trial period (females only)
* Refrain from blood donation during the trial
* Give written informed consent
* Allow the Investigator to register volunteer details with a confidential database (The Over-volunteering Protection Service) to prevent concurrent entry into clinical trials
* Able and willing (in the Investigator's opinion) to comply with all the trial requirements

Exclusion Criteria:

Volunteers must meet none of the following criteria to enter the trial:

* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the trial period
* Prior vaccination with candidate vaccine MVA85A, candidate vaccine FP85A,any other recombinant MVA vaccine or any other candidate TB vaccine
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned trial vaccination date
* Clinically significant history of skin disorder, allergy, atopy, immunodeficiency (including HIV), cancer (except BCC or CIS), cardiovascular disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder, neurological illness, psychiatric disorder, drug or alcohol abuse
* Concurrent oral or systemic steroid medication or the concurrent use of other immunosuppressive agents
* History of anaphylaxis to vaccination or any allergy likely to be exacerbated by any component of the trial vaccine, sedative drugs, or any local or general anaesthetic agents
* Pregnancy, lactation or intention to become pregnant during trial period
* Any respiratory disease, including asthma
* Current smoker
* Clinically significant abnormality on screening CT thorax
* Clinically significant abnormality of pulmonary function tests
* Any nasal, pharyngeal, or laryngeal finding which precludes bronchoscopy
* Current use of any medication taken through the nasal or inhaled route including cocaine or other recreational drugs
* Clinical, radiological, or laboratory evidence of current active TB disease
* Past treatment for TB disease
* Any clinically significant abnormality of screening blood or urine tests
* Positive HBsAg, HCV or HIV antibodies
* Any other significant disease, disorder, or finding, which, in the opinion of the Investigator, may either put the volunteer at risk, affect the volunteer's ability to participate in the trial or impair interpretation of the trial data

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2015-09; Primary Completion 2018-10-04 (Actual); Study Completion 2018-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen McShane, Study Director — University of Oxford; Paul Moss, Principal Investigator — University of Birmingham; Marc Lipman, Principal Investigator — Royal Free Hostpital; Felicity Perrin, Principal Investigator — King's College Hospital NHS Trust
Locations (5):
- United Kingdom (5):
  - Centre for Clinical Vaccinology and Tropical Medicine (CCVTM), Churchill Hospital, Oxford, Oxfordshire
  - John Warin Ward, Churchill Hospital, Oxford, Oxfordshire
  - NIHR Wellcome Trust Clinical Research Facility, University of Birmingham, Birmingham, West Midlands
  - NIHR/Wellcome Trust King's Clinical Research Facility, London
  - Royal Free Hospital NHS Foundation Trust, London

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Receive 5x10^7 pfu aerosol inhaled MVA85A
Period: Overall Study
Arm/Group | Starter Group | Group A
Started | 2 | 0
Completed | 2 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Starter Group: Received 1x10^7 pfu aerosol inhaled MVA85A at day 0.
Arm/Group | Starter Group
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 2

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events (AE)
Description: Actively and passively collected data on adverse events via diary card for 14 days after vaccination and at each visit over 6 months.
Time Frame: Up to Day 168
Measure: Count of Participants; unit: Participants
Groups:
- Starter Group: Receive 1x10^7 pfu aerosol inhaled MVA85.
Arm/Group | Starter Group
Number analyzed (Participants) | 2
Participants | 2

2. Secondary Outcome: Laboratory Markers of Immunity
Description: Evaluation of ex-vivo ELISpot and intracellular cytokine staining in blood and bronchoalveolar lavage (BAL) samples.
Time Frame: Up to Day 168
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All AEs occurring for 6 months following the vaccination that were observed by the investigator or reported by the volunteer, whether or not attributed to study medication, were recorded by volunteers on electronic diary cards or by staff on CRFs.
Arm/Group | Starter Group
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Starter Group (N=2)
radiological changes (Investigations) | 1 (1) — transient asymptomatic radiological changes to the lung on CT scan at Day 28.

LIMITATIONS AND CAVEATS:
Due to significant challenges with recruitment at all UK sites this study has been terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-19): https://cdn.clinicaltrials.gov/large-docs/36/NCT02532036/Prot_SAP_000.pdf